CLINICAL TRIAL: NCT07109960
Title: Effect of Isometric Exercise Versus Hand Reflexology on Hemodynamic Parameters, Fatigue, and Anxiety Among Patients With Acute Myocardial Infarction: A Randomized Clinical Trial
Brief Title: Effect of Isometric Exercise Versus Hand Reflexology on Hemodynamic Parameters Among Patients With AMI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Bahaa Mirza Skal, Lecturer, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: bahaa198811
Record Dates: First submitted 2025-07-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Hemodynamic Parameters; Fatigue; Anxiety
Keywords: Isometric Exercise; Hand Reflexology; Acute Myocardial Infarction
MeSH Terms: conditions — Fatigue; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Each participant in the isometric exercise group receives included ankle exercises, knee workouts, head exercises, static abdominis exercises, and sustained hand grip exercises. Every contraction lasted for 10 seconds, 10 repetitions, two IE sessions over a period of three days. Each IE session lasted between 25 and 35 minutes.
  Each participant in the hand reflexology group underwent two the sessions of hand reflexology. Each session had a duration of 15 minutes, which was then followed by a five-minute period of rest.
  While isometric exercise- hand reflexology experimental group was given for the participant, the same intervention of isometric exercise and hand reflexology groups Furthermore, no interventions were done for the control group (received routine care only).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric exercise, hand reflexology, isometric exercise-hand reflexology, and control groups (Experimental): Each participant in the isometric exercise group receives included ankle exercises, knee workouts, head exercises, static abdominis exercises, and sustained hand grip exercises. Every contraction lasted for 10 seconds, 10 repetitions, two IE sessions over a period of three days. Each IE session lasted between 25 and 35 minutes. Each participant in the hand reflexology group underwent two the sessions of hand reflexology. Each session had a duration of 15 minutes, which was then followed by a five-minute period of rest. While isometric exercise- hand reflexology experimental group was given for the participant, the same intervention of isometric exercise and hand reflexology groups.
  Interventions: Other: Isometric exercise and hand reflexology
- Routine care (No Intervention): no interventions were done for the control group (received routine care only).

INTERVENTIONS:
Other: Isometric exercise and hand reflexology — Each participant in the isometric exercise group receives included ankle exercises, knee workouts, head exercises, static abdominis exercises, and sustained hand grip exercises. Every contraction lasted for 10 seconds, 10 repetitions, two IE sessions over a period of three days. Each IE session lasted between 25 and 35 minutes.
  Each participant in the hand reflexology group underwent two the sessions of hand reflexology. Each session had a duration of 15 minutes, which was then followed by a five-minute period of rest.
  While isometric exercise- hand reflexology experimental group was given for the participant, the same intervention of isometric exercise and hand reflexology groups Furthermore, no interventions were done for the control group (received routine care only).
  Arms: Isometric exercise, hand reflexology, isometric exercise-hand reflexology, and control groups

SUMMARY:
The goal of this clinical trial is to evaluate the comparative effect of isometric exercise versus hand reflexology on primary hemodynamic parameters, fatigue, and anxiety in patients with acute myocardial infarction.

Researcher will know which one of the interventional procedures (isometric exercise, hand reflexology, or hand reflexology and hand reflexology) was more effective to primary hemodynamic parameters, fatigue, and anxiety.

Each participant in the isometric exercise group receives included ankle exercises, knee workouts, head exercises, static abdominis exercises, and sustained hand grip exercises. Every contraction lasted for 10 seconds, 10 repetitions, two IE sessions over a period of three days. Each IE session lasted between 25 and 35 minutes.

Each participant in the hand reflexology group underwent two the sessions of hand reflexology. Each session had a duration of 15 minutes, which was then followed by a five-minute period of rest

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) encompass a group of medical conditions including angina pectoris, myocardial infarction, congestive heart failure, irregular rhythms, cardiac valve disease, and aortic atherosclerosis. Clinical CVD is the accumulation of plaque in the arteries that provide blood to the cardiac muscle. Plaque-clogged arteries undergo hardening, resulting in reduced blood flow through them. The specific site of the plaque dictates the type of cardiac defect.

Whenever there is a need to improve patient symptoms or prognosis by obtaining information about the severity through disease of coronary artery, it is recommended to use the invasive coronary angiography (ICA). The femoral artery area commonly experiences various local vascular complications, including minor or major bleeding, hematoma, pseudoaneurysm, and arteriovenous (AV) fistula. These complications arise due to the frequent use of the femoral artery for vascular access procedures.

Cardiac patients typically exhibit a higher prevalence of anxiety compared to people with other medical conditions. Approximately 80% of individuals with cardiac conditions are reported to exhibit and manifest anxiety before to cardiac arrest. The primary factors contributing to patient anxiety include previous encounters, discomfort, emotional strain, unfamiliar environments.

An acute myocardial infarction (AMI) occurs due to decreased blood flow inside the coronary arteries. Ischemia and myocardial damage may an elevating or descending ST segment on the Electrocardiogram (ECG). Among the consequences of AMI include arrhythmia and alterations in physiological parameters including hypertension, hypotension, tachypnea, and fever.

Isometric exercise occurs a feature pressor rase in blood flow which may significant in keep provide of muscle through continuous contraction. the response is middle by joint central and peripheral occur input to the medullary of cardiovascular the centers. In the normal persons the rise in blood flow is middle through a increase in output of heart with no change in resistance of systemic vascular.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: Adults aged 18 to 75 years.
2. Confirmed diagnosis of acute myocardial infarction (AMI).
3. Time since AMI.
4. Stable clinical condition.
5. Informed consent.
6. No contraindications to interventions (severe musculoskeletal or neurological impairments).
7. No current use of reflexology.
8. No recent cardiovascular surgery.
9. No uncontrolled co-morbidities such as DM, COPD, or chronic kidney disease.
10. Stable medication regimen within the past 24 hours.
11. No severe psychological disorders (e.g., major depressive disorder, schizophrenia).
12. Ability to complete study protocol.

Exclusion Criteria:

1. Severe or ongoing cardiovascular events.
2. Heart failure.
3. Severe renal or hepatic impairment.
4. Active or uncontrolled infections.
5. Major surgical intervention.
6. Severe musculoskeletal, neurological disorders.
7. Severe psychiatric disorders.
8. Current participation in other interventional trials.
9. Pregnancy or lactation.
10. Inability to follow protocol.
11. Significant uncontrolled comorbidities (HTN, DM).
12. Known allergy to reflexology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Patients' blood pressure were measured and recorded 15 minutes before intervention by researcher, and 15 minutes after the completion of intervention
  Blood pressure (right hand lying on the back) was measured through digital blood pressure monitor (RossMax MG150f, made in Tiwan).
Fatigue | Patients' fatigue were measured and recorded 15 minutes before intervention by patient, and 15 minutes after the completion of intervention
  Fatigue visual analogue scale (VAS) was used to measure fatigue. VAS is a self-administered visual scale that includes a 10 cm horizontal line graded from 0 to 10. Zero indicates no fatigue, 1-3 indicates mild fatigue, 4-7 indicates moderate fatigue, and 8-10 indicates severe fatigue.
Anxiety | Patients' fatigue were measured and recorded 15 minutes before intervention by patient, and 15 minutes after the completion of intervention
  State- Trait Anxiety Inventory (STAI) is a reliable and valid instrument that was developed by Spielberger in 1983 with a range of internal consistency coefficients from 0.86- 0.95.

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa M Skal, PhD, Principal Investigator — Qadisiyah University-Faculty of Nursing
Locations (1):
- Al-Diwaniyah government hospital, Al Qādisīyah, AL-Diwaniya, Iraq

IPD SHARING:
Plan to Share IPD: No